CLINICAL TRIAL: NCT03113474
Title: Profiling the Endocannabinoid Response to Hedonic Eating
Acronym: Lekkere trek
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL51830.081.14
Record Dates: First submitted 2017-04-09; First posted 2017-04-13 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Obesity; Food Preferences
MeSH Terms: conditions — Obesity; Food Preferences

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palatable-neutral (Experimental): Participants are exposed to palatable food in the first test session, and to the neutral food in the second test session.
  Interventions: Other: Food palatability
- Neutral-palatable (Experimental): Participants are exposed to neutral food in the first test session, and to the palatable food in the second test session.
  Interventions: Other: Food palatability

INTERVENTIONS:
Other: Food palatability — Food palatability is modulated

SUMMARY:
Study into the endocannabinoid response to consuming a palatable versus a neutral food.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (self-report)
* Dutch
* Evaluating one of the used foods as palatable
* Evaluating one of the used foods as neutral
* Hb value between 8.1 and 11.0 mmol/L at screening

Exclusion Criteria:

* restraint eating
* lack of appetite
* difficulties eating/swallowing
* endocrine disorders
* energy restricted diet two months prior to study
* weight change > 5 kg in two months prior to study
* stomach or bowel disease
* taste or smell disorders (self-report)
* not consuming foods used in the study
* smoking > 1 cigarette per day
* drinking > 21 units alcohol per week

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2015-10-08 (Actual); Study Completion 2015-10-08 (Actual)

PRIMARY OUTCOMES:
Endocannainoid levels | prior to, during and two hours after eating
  To assess changes in endocannabinoid plasma levels prior to, during and after eating a palatable versus a neutral food

SECONDARY OUTCOMES:
Pancreatic polypeptide (pg/ml) | prior to, during and two hours after eating
  To assess changes in pancreatic polypeptide plasma levels prior to, during and after eating a palatable versus a neutral food
Ghrelin (pg/ml) | prior to, during and two hours after eating
  To assess changes in ghrelin plasma levels prior to, during and after eating a palatable versus a neutral food

IPD SHARING:
Plan to Share IPD: Undecided